CLINICAL TRIAL: NCT02566798
Title: Anti-inflammatory Effect of Serum of Osteoarthritis Patients After Administration of the Oléogrape®SEED, an Extract of Grape and Olive
Acronym: OléograpeSEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RC15_0173
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oleogrape (Experimental): Patients are taking capsules of OleograpeSEED (Extract of grape and olive) 3 times a day (1mg/day) in the morning, at noon and in the evening during 7 days
  Interventions: Drug: Extract of grape and olive
- Placebo (Placebo Comparator): Patients are taking capsules of placebo (lactose) 3 times a day in the morning, at noon and in the evening during 7 days
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: Extract of grape and olive — Patients are taking capsules of OleograpeSEED 3 times a day (1mg/day) in the morning, at noon and in the evening during 7 days.
  Blood samples and synovial fluid are performed on D0 and D7
  Other Names: OleograpeSEED
  Arms: Oleogrape
Drug: Lactose — Patients are taking capsules of placebo 3 times a day in the morning, at noon and in the evening during 7 days.
  Blood samples and synovial fluid are performed on D0 and D7
  Arms: Placebo

SUMMARY:
Osteoarthritis is a degenerative disease that affects a growing proportion of the population. There is currently no treatment to halt this process. The aim of the research is in particular to find treatments targeting the molecular origins of osteoarthritis focusing especially on the inflammatory component of the disease. That is why research is looking to the development of preventive treatments like nutraceuticals. This project aims to determine the anti-inflammatory properties of sera of patients who received supplementation of their diet with an extract of grape and olive: the Oléogrape®SEED. Sera and synovial fluid will be collected during visits for hyaluronic acid injections in OA patients. These sera will be tested in vitro in a model of inflamed chondrocytes.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old and over
* Patients with knee osteoarthritis (ACR criteria)
* Patients requiring injection of hyaluronic acid (no corticosteroid associated)
* Radiological stage of knee osteoarthritis 1, 2 or 3 (Kellgren-Lawrence)
* Informed consent form signed

Exclusion Criteria:

* younger than 50 years
* protected adult
* Pregnant woman
* Radiological Stage 4 osteoarthritis (Kellgren-Lawrence)
* knee osteoarthritis secondary to arthritis
* Taking a long term treatment of osteoarthritis (Piasclédine®, Diacéréine®, glucosamine, chondroitin)
* inflammatory pathology other than osteoarthritis
* Taking anti-inflammatory medications
* Refusal to participate in the study
* Use of food supplements with anti-inflammatory properties
* Arthroscopy less than 6 months
* corticosteroid injection <3 months
* INR> 4 or TCA> 2 (anticoagulants)
* Being allergic to lactose

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
biochemical assays of NO production in the cell culture supernatant to measure the anti-inflammatory action of patients' sera | 7 days
biochemical assays of PGE2 production in the cell culture supernatant to measure the anti-inflammatory action of patients' sera | 7 days

SECONDARY OUTCOMES:
qualitative evaluation by mass spectrometry to assess the bioavailability of polyphenols in the patients' sera | 7 days